CLINICAL TRIAL: NCT00959530
Title: A Randomized Clinical Trial Comparing Lingualized and Full Bilaterally Balanced Articulation for Complete Dentures
Brief Title: Comparison of Lingualized and Full Bilaterally Balanced Articulation
Acronym: denture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nihon University (Other)
Responsible Party: Principal Investigator, Yasuhiko Kawai, Professor, Nihon University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07-014
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Jaw, Edentulous
Keywords: complete dentures; patient satisfaction; treatment cost
MeSH Terms: conditions — Jaw, Edentulous; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- lingualized (Experimental): complete denture fabricated by lingualized occlusion scheme
  Interventions: Procedure: lingualized occlusion
- Full Bilaterally Balanced Articulation (Placebo Comparator): complete denture fabricated by Full Bilaterally Balanced Articulation scheme
  Interventions: Procedure: Full Bilaterally Balanced Articulation

INTERVENTIONS:
Procedure: lingualized occlusion — occlusal surface arranged by lingualized occlusion
  Other Names: e-ha artificial teeth, shofu porcelain teeth
  Arms: lingualized
Procedure: Full Bilaterally Balanced Articulation — occlusal surface arranged by Full Bilaterally Balanced Articulation
  Other Names: Shofu Ace Posterior
  Arms: Full Bilaterally Balanced Articulation

SUMMARY:
The purpose of this study is to find the difference between patient satisfaction, masticatory performance and cost between two occlusal schemes for complete denture prosthodontics.

DETAILED DESCRIPTION:
Two occlusal scheme applied to complete denture prosthodontics has been compared in RCT. This will have clinical benefit for deciding which occlusal scheme is better according to patient conditions. It will also have impact on dental educational curriculum.

ELIGIBILITY:
Inclusion Criteria:

* edentulous both maxilla and mandible, asking for new denture fabrication

Exclusion Criteria:

* psychiatric problem
* those who have difficulty answering the questionnaire
* oral cancer
* radiation experience

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-11; Primary Completion 2009-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
patient satisfaction on 100mm visual analogue scale | 6month

SECONDARY OUTCOMES:
treatment cost | 6month

CONTACTS AND LOCATIONS:
Overall Officials: Yasuhiko Kawai, DDS MMedSc, Principal Investigator — Nihon University; Yuichi Matsumaru, DDS, Principal Investigator — Nihon University
Locations (1):
- Nihon University Hospital, Matsudo, Chiba, Japan

REFERENCES:
- [Background] Heydecke G, Vogeler M, Wolkewitz M, Turp JC, Strub JR. Simplified versus comprehensive fabrication of complete dentures: patient ratings of denture satisfaction from a randomized crossover trial. Quintessence Int. 2008 Feb;39(2):107-16. PMID 18560649
- [Background] Sutton AF, Worthington HV, McCord JF. RCT comparing posterior occlusal forms for complete dentures. J Dent Res. 2007 Jul;86(7):651-5. doi: 10.1177/154405910708600713. PMID 17586713
- [Background] Sutton AF, McCord JF. A randomized clinical trial comparing anatomic, lingualized, and zero-degree posterior occlusal forms for complete dentures. J Prosthet Dent. 2007 May;97(5):292-8. doi: 10.1016/j.prosdent.2007.03.003. PMID 17547948
- [Background] Kimoto S, Gunji A, Yamakawa A, Ajiro H, Kanno K, Shinomiya M, Kawai Y, Kawara M, Kobayashi K. Prospective clinical trial comparing lingualized occlusion to bilateral balanced occlusion in complete dentures: a pilot study. Int J Prosthodont. 2006 Jan-Feb;19(1):103-9. PMID 16479769
- [Derived] Matsumaru Y. Influence of mandibular residual ridge resorption on objective masticatory measures of lingualized and fully bilateral balanced denture articulation. J Prosthodont Res. 2010 Jul;54(3):112-8. doi: 10.1016/j.jpor.2009.11.008. Epub 2010 Jan 19. PMID 20089469